CLINICAL TRIAL: NCT03572010
Title: A Novel Stable Iron Isotope Method to Define Iron Needs and Improve Iron Nutrition in HIV+ and HIV- Children
Brief Title: Stable Iron Isotope Method in HIV+ and HIV- Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Fe_HIV
Record Dates: First submitted 2018-05-16; First posted 2018-06-28 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FeFum fortified maize test meal (Placebo Comparator)
  Interventions: Dietary Supplement: FeFum fortified maize test meal
- FeSO4 fortified LNS (Placebo Comparator)
  Interventions: Dietary Supplement: FeSO4 fortified LNS
- FeSO4 supplement (Placebo Comparator)
  Interventions: Dietary Supplement: FeSO4 supplement
- FeSO4 fortified fruit juice (Placebo Comparator)
  Interventions: Dietary Supplement: FeSO4 fortified fruit juice

INTERVENTIONS:
Dietary Supplement: FeFum fortified maize test meal — Maize porridge extrinsically labeled with 2 mg ferrous fumarate (58FeFum); only for iron deficient children (defined by plasma ferritin <40 mikrogramm/L and/or sTfR >8.3 mg/L); cereal staple foods, like maize, depending on milling, may be high in phytic acid, a potent iron absorption inhibitor
  Arms: FeFum fortified maize test meal
Dietary Supplement: FeSO4 fortified LNS — self-made Lipid-based nutritional supplement (LNS) extrinsically fortified and labeled with 6 mg ferrous sulfate (57FeSO4); only for iron deficient children (defined by plasma ferritin <40 mikrogramm/L and/or sTfR >8.3 mg/L); LNS may be a better food matrix for iron supplementation compared to maize-based porridge; contains canola oil, peanut paste, milk powder, sugar, maltodextrin and palm stearin
  Arms: FeSO4 fortified LNS
Dietary Supplement: FeSO4 supplement — 170 mg iron tablets as FeSO4 (containing 55 mg of elemental iron) with 6 mg extrinsically labeled 57Fe; will be given together with a glass of water; only for iron deficient children (defined by plasma ferritin <40 mikrogramm/L and/or sTfR >8.3 mg/L);
  Arms: FeSO4 supplement
Dietary Supplement: FeSO4 fortified fruit juice — Fruit juice labeled with 12 mg 57Fe as FeSO4; in the group for iron sufficient children
  Arms: FeSO4 fortified fruit juice

SUMMARY:
The objective of this study is to compare HIV infected children to uninfected children regarding 1) quantifying iron absorption from iron fortified maize porridge, lipid-based food supplements and oral iron supplements, and 2) quantifying the daily iron requirement.

DETAILED DESCRIPTION:
In Sub-Saharan Africa, HIV is a major cause of morbidity and mortality in children. Anemia frequently complicates pediatric HIV infection and predicts disease progression and mortality. Iron requirements and the specific contribution of iron deficiency (ID) to anemia in pediatric HIV infection remains uncertain. The fundamental barrier to understanding iron nutrition in HIV infection is that sub-clinical inflammation in individuals with HIV infection confounds the usual bio-markers used to assess iron status and response to iron interventions. A novel iron stable isotope technique developed by ETH Zurich, Switzerland, is a promising new tool for better understanding of iron metabolism in HIV infection. In contrast to existing conventional bio-markers of iron status, a method based on isotopic dilution of whole body iron labeled with stable, non-radioactive isotopes of iron (58Fe, 57Fe) could directly quantify iron requirements, as well as iron absorption from interventions, completely free of bias and confounding by inflammation. This method could offer, for the first time, a long-term quantitative measure of iron balance and absorption from iron interventions and provide reliable data on which to base nutrition recommendations for HIV infection.

The objective is to compare HIV infected children to uninfected children: 1) Quantify iron absorption from iron fortified maize porridge, lipid-based food supplements and oral iron supplements; 2) Quantify the daily iron requirement.

The study participants will be recruited from the South African Stellenbosch University/Tygerberg Children's Hospital long-term antiretroviral therapy (ART) cohort of perinatally HIV infected children and uninfected controls from the same communities, matched by age and gender. As a secondary outcome, we want to investigate the effect of iron supplementation on the gut microbiome.

In study 1, using a randomized cross-over design and stable isotope labeled single meal/doses the investigators will: a) quantify the impairment of dietary iron absorption in HIV infected, iron deficient children compared to HIV uninfected, iron deficient controls using a labeled iron fortified maize meal, a lipid-based nutritional supplement (LNS) and an oral iron supplement; and b) administer sufficient iron isotope label (57Fe) to allow equilibration and follow up of isotopic composition in the blood for two years (isotope dilution technique). At the end of Study 1, all iron deficient children will be iron replete prior to entering Study 2. In study 1, in parallel, a group of HIV infected and uninfected, iron sufficient children will be given orally 12 mg 57Fe as ferrous sulfate (FeSO4).

In study 2, the investigators will apply the principle of long-term isotope dilution to quantify the daily iron requirement in both the HIV infected and uninfected children, and the difference in iron requirements.

The overall goal is to provide optimized recommendations on dietary iron requirements and iron treatment regimens in HIV infected children, in order to reduce ID and anemia, improve their health and well-being, their long-term prognosis and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-13 years at baseline
* Hemoglobin >=8 g/dL
* BMI -3 to 3 SD of reference population
* HIV criteria: soluble cluster of differentiation 4 (sCD4) >=500 cells/mm^3, HIV RNA viral load <50 copies/mL (measured as part of routine care)
* Plasma ferritin <30 mikrogramm/L
* The caregiver is willing to participate in the study
* The caregiver speaks English, Afrikaans or isiXhosa
* The informed consent form has been read and signed by the caregiver (or has been read out to the caregiver in case of illiteracy) plus assent needs to be obtained from the child
* Residence in the study site for the period of the study.

For non-iron deficient children:

* Hemoglobin >=11.5 g/dL
* Plasma ferritin >=40 mikrogramm/L

Exclusion Criteria:

* Iron supplements 3 months prior to study start
* Food allergy or intolerance against peanuts or milk
* Acute illness or other conditions that in the opinion of the PI or co-researchers would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Participants taking part in other studies requiring the drawing of blood
* Not planning long-term residence in study site.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption | Measured 14 days after consumption of the 3 different types of iron vehicles (Days 17 and 31); Enrichment shift of iron isotopes into red blood cells from Day 31 to 451
  Iron absorption will be measured from the 3 different types of iron vehicles from the iron deficient group (FeFum fortified maize porridge, FeSO4 containing LNS, FeSO4 supplement). It is estimated that iron absorption is lower in HIV infected children.

SECONDARY OUTCOMES:
Hemoglobin in g/dL (in blood) | Days -1, 17 (in iron deficient children), 31, 151, 271, 361, 451
  to identify anemia
Plasma ferritin in µg/L (in blood) | Days -1, 17 (in iron deficient children), 31, 151, 271, 361, 451
  to identify iron deficiency
Soluble transferrin receptor in mg/L (in blood) | Days -1, 17 (in iron deficient children), 31, 151, 271, 361, 451
  to identify iron deficiency
Transferrin saturation in % (in blood) | Days -1, 17 (in iron deficient children), 31, 151, 271, 361, 451
  to calculate percent of transferrin that has iron bound to it; Plasma iron and transferrin saturation will be combined to calculate transferrin saturation (ratio)
Erythropoetin (in blood) | Days -1, 17 (in iron deficient children), 31, 151, 271, 361, 451
  produced in kidney and triggers production of red blood cells
C-reactive protein in mg/L (in blood) | Days -1, 17 (in iron deficient children), 31, 151, 271, 361, 451
  to identify acute inflammation, which inhibits iron absorption
alpha-1-glycoprotein in g/L (in blood) | Days -1, 17 (in iron deficient children), 31, 151, 271, 361, 451
  to identify chronic inflammation, which inhibits iron absorption
Plasma hepcidin (in blood) | Days -1, 17 (in iron deficient children), 31, 151, 271, 361, 451
  one of major iron absorption regulators
Interleukin-6 (in blood) | Days -1, 17 (in iron deficient children), 31, 151, 271, 361, 451
  systemic inflammation marker
Intestinal fatty acid binding protein 1 and 2 (in blood) | Days -1, 17 (in iron deficient children), 31, 151, 271, 361, 451
  inflammation marker for gut integrity
Lipopolysaccharide binding protein (in blood) | Days -1, 17 (in iron deficient children), 31, 151, 271, 361, 451
  immune response marker
Fecal calprotectin (in stool) | Days -1, 31 and 121 (in iron deficient children)
  gut inflammation marker

CONTACTS AND LOCATIONS:
Locations (1):
- Familiy Clinical Research Unit (FAMCRU), Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goosen C, Proost S, Baumgartner J, Mallick K, Tito RY, Barnabas SL, Cotton MF, Zimmermann MB, Raes J, Blaauw R. Associations of HIV and iron status with gut microbiota composition, gut inflammation and gut integrity in South African school-age children: a two-way factorial case-control study. J Hum Nutr Diet. 2023 Jun;36(3):819-832. doi: 10.1111/jhn.13171. Epub 2023 Apr 16. PMID 36992541
- [Derived] Goosen C, Proost S, Tito RY, Baumgartner J, Barnabas SL, Cotton MF, Zimmermann MB, Raes J, Blaauw R. The effect of oral iron supplementation on the gut microbiota, gut inflammation, and iron status in iron-depleted South African school-age children with virally suppressed HIV and without HIV. Eur J Nutr. 2022 Jun;61(4):2067-2078. doi: 10.1007/s00394-021-02793-9. Epub 2022 Jan 8. PMID 34997267
- [Derived] Goosen C, Baumgartner J, Mikulic N, Barnabas SL, Cotton MF, Zimmermann MB, Blaauw R. Examining Associations of HIV and Iron Status with Nutritional and Inflammatory Status, Anemia, and Dietary Intake in South African Schoolchildren. Nutrients. 2021 Mar 16;13(3):962. doi: 10.3390/nu13030962. PMID 33809705